CLINICAL TRIAL: NCT00005117
Title: Effect of Pravastatin on Endothelial Dysfunction Following a Single High Fat Meal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00051-1162; M01RR000051 (NIH)
Record Dates: First submitted 2000-04-18; First posted 2000-04-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Heart Diseases
Keywords: endothelial dysfunction
MeSH Terms: conditions — Heart Diseases | interventions — Pravastatin

INTERVENTIONS:
Drug: pravastatin

SUMMARY:
There is significant evidence that HMG-CoA reductase inhibitors, a commonly used class of cholesterol lowering medications, reduce the risk of death from coronary disease. Although these medicines lower cholesterol levels, other studies suggest that they have an additional effect on improving blood vessel functioning. It has also been shown that consumption of a fatty meal temporarily alters blood vessel functioning, causing endothelial dysfunction. This study will examine if pravastatin, an HMG-CoA reductase inhibitor, improves blood vessel functioning after a fatty meal. We plan on enrolling 32 subjects, aged 18-40 years, who are healthy with no history of diabetes, smoking, high blood pressure, or heart disease. These subjects will be randomly assigned to initially receive four days of pravastatin or an inactive substance, and then crossed over to the other group. Blood vessel functioning will be monitored by a technique called flow mediated vasoactivity, which uses ultrasound measurement of the forearm artery and its response to temporary occlusion. This primary measure of flow mediated vasoactivity will be done before and after consumption of a fatty meal. We hope to show that treatment with pravastatin prevents the blood vessel dysfunction known to occur after a high fat meal. Secondary outcomes will include measurement of endothelin-l, a mediator of blood vessel functioning, and assessment of changes in lipid profiles. If pravastatin does prevent endothelial dysfunction in this setting, it could lead to further studies about their use in more acute medical settings, including heart attacks or strokes.

ELIGIBILITY:
Inclusion Criteria:

* No history of the following: hypertension, diabetes mellitus, smoking, and coronary artery disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 4200 E. 9th Avenue, Box B133, Denver, Colorado, United States